CLINICAL TRIAL: NCT01422902
Title: Evaluation of a Cognitive Adaptive E-treatment in Schizophrenia-diagnosed Adults, A Remediation-based Approach
Brief Title: Evaluation of a Cognitive Adaptive E-treatment in Schizophrenia-diagnosed Adults
Acronym: e-CAeSAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Posit Science Corporation (Industry)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BPI-1001-11; IRC2MH909833-01 (Other Grant/Funding Number: National Institutes of Mental Health)
Record Dates: First submitted 2011-08-22; First posted 2011-08-25 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Cognitive deficits; Cognitive remediation; Software; Brain Plasticity
MeSH Terms: conditions — Schizophrenia; Cognition Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Plasticity-based Cognitive Training (Experimental): Computerized plasticity-based adaptive cognitive training, up to 130 hours
  Interventions: Other: Plasticity-based Cognitive Training
- Non-plasticity-based Training (Active Comparator): Commercially available computerized training, up to 130 hours
  Interventions: Other: Non-plasticity-based Training

INTERVENTIONS:
Other: Plasticity-based Cognitive Training
  Other Names: brainhq
  Arms: Plasticity-based Cognitive Training
Other: Non-plasticity-based Training — Computer games
  Arms: Non-plasticity-based Training

SUMMARY:
This study is a multi-site, double-blind, randomized, controlled clinical trial to assess the safety and effectiveness of plasticity-based, adaptive, computerized-based cognitive remediation treatment versus a computer-based control.

The investigators proposed that a computerized cognitive remediation program based upon the principles of brain plasticity may improve information processing and thus drive clinically significant improvements in cognitive and functional performance in individuals with schizophrenia.

DETAILED DESCRIPTION:
The symptoms of schizophrenia fall into three main categories: positive symptoms, negative symptoms, and cognitive symptoms. Each category represents distinct functional challenges and impedes patient productivity and overall quality of life.

Cognitive symptoms are pervasive and result in deficits in executive functioning (the ability to understand information and use it to make decisions), attention (the ability to identify, select, and focus on relevant sensory events), and working memory (the ability to hold information in memory and then guide actions from it). These symptoms impair patients' abilities to successfully perform everyday activities, including independent living, employment, and social relationships, and in addition can cause great emotional distress.

Cognitive impairment in schizophrenia has now received substantial academic study, with over 24,000 research papers published in the field since 1990. This enormous body of work has shown that cognitive impairment is likely to be present in virtually all patients with schizophrenia, regardless of their severity of illness or treatment status. People with schizophrenia typically perform 1-2 standard deviations below the mean of age-matched controls (indicating substantial impairment) across the domains of speed of information processing, attention, working memory, verbal and visual learning, reasoning and social cognition.

While cognitive impairment in schizophrenia was originally assumed to be secondary to positive or negative symptoms of the disorder, or related to the use of anti-psychotic medications, recent research has conclusively shown that neither of these past assumptions is true. For example, the landmark Clinical Antipsychotic Trials of Intervention Effectiveness (CATIE) trial involving 1,493 participants demonstrated that negative symptoms are only mildly correlated with cognitive function, and that positive symptoms are completely uncorrelated with cognitive function. Furthermore, research has shown that cognitive impairment is evident in people with schizophrenia before they are medicated, prior to diagnosis, and in first-degree relatives of people diagnosed with schizophrenia; indicating that medication is not the cause of cognitive impairment. In aggregate, these data have established the well-accepted current viewpoint that cognitive dysfunction is a core primary symptom and deficit in schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of older with confirmed diagnosis of Schizophrenia
* Adequate decisional and reading capacity
* Clinical stable
* Moderate or less severity on Positive and Negative Symptoms Scale
* English speaker
* Capable of completing clinical and cognitive assessment battery
* Lack of visual, auditory or motor capacity to participate in the study
* Minimal level of extrapyramidal symptoms
* Minimal level of depressive symptoms

Exclusion Criteria:

* Failure to meet suicidality rating criteria
* Prescribed greater than 2 anti-psychotics
* Significant alcohol and illicit drug use
* History of mental retardation or pervasive developmental disorder or other neurological disorder
* Prior specified computer-based cognitive remediation training
* Participation in a concurrent study that could affect the outcome of this one

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-04; Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of the effects of plasticity-based, adaptive cognitive remediation on cognitive abilities, functional status and quality of life. | 6 Months
  Each outcome score (MCCB composite score and UPSA-2 total score) will be analyzed separately. The treatment efficacy will be established if and only if both tests on MCCB and UPSA-2 are significant at two-sided alpha level of 0.05.

SECONDARY OUTCOMES:
Demonstration of equivalency in safety effects reported between treatment groups. | 6 Months
  Positive and Negative Symptom Scale (PANSS) positive symptom scale, negative symptom scale and total scale will be assessed at study mid-point and study end. Adverse effects by treatment group will also be assessed at study mid-point and study end.

CONTACTS AND LOCATIONS:
Overall Officials: Henry W. Mahncke, PhD, Principal Investigator — Posit Science Corporation; Richard Keefe, PhD, Principal Investigator — Schizophrenia Trials Network; Scott Stroup, MD, MPH, Principal Investigator — Schizophrenia Trials Network; Cate Stasio, Study Director — Posit Science Corporation
Locations (2):
- United States (2):
  - Palo Alto Veteran's Affairs Medical Center, Palo Alto, California
  - Posit Science Corporation, San Francisco, California